CLINICAL TRIAL: NCT06563349
Title: The Effect of Intravenous Magnesium Infusion on the Opioid Consumption, the Circulatory, Metabolic and Hormonal Response to Intubation and Surgical Trauma During Anaesthesia for Laparoscopy in Children. Randomized Clinical Trial.
Brief Title: Magnesium Sulfate in Children Undergoing Laparoscopic Appendectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Maciej Kaszyński, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Mg01
Record Dates: First submitted 2024-08-05; First posted 2024-08-20 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Opioid Consumption; Multimodal Analgesia; Acute Appendicitis; Complication of Treatment
Keywords: multimodal analgesia; magnesium sulfate; laparoscopic appendectomy; children; pediatric population; adjuvant; metabolic stress response; hormonal response; inflammatory response
MeSH Terms: conditions — Appendicitis | interventions — Intravital Microscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drug or placebo (normal saline) will be placed in a syringe by the principal investigator. Only principal investigator will be aware of the participants allocation. The principal investigator will not be involved in the process of: recruitment, providing an intervention, or outcomes assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulfate (Experimental): 10% magnesium sulfate intravenous bolus of 0.5 ml/kg (maximum 20 ml) over 5 min before induction of anesthesia followed by magnesium sulfate infusion at 0.15 ml/kg/h (maximum 6 ml/h) intraoperatively will be administered. The infusion will be discontinued before the patients' transfer to the postanesthesia care unit.
  Interventions: Drug: Intravenous magnesium sulfate
- Control (Placebo Comparator): 0.9% NaCl (sodium chloride) intravenous bolus of 0.5 ml/kg (maximum 20 ml) over 5 min before induction of anesthesia followed by 0.9% NaCl infusion at 0.15 ml/kg/h (maximum 5ml/h) intraoperatively will be administered. The infusion will be discontinued before the patients' transfer to the postanesthesia care unit.
  Interventions: Drug: Normal saline infusion

INTERVENTIONS:
Drug: Intravenous magnesium sulfate — Intraoperative intravenous magnesium sulfate infusion.
  Other Names: IVM (intravenous magnesium)
  Arms: Magnesium Sulfate
Drug: Normal saline infusion — Intraoperative intravenous normal saline infusion.
  Other Names: Placebo
  Arms: Control

SUMMARY:
Magnesium sulfate is one of the most commonly used co-analgetics. Its antinociceptive effect is related to antagonizing NMDA (N-methyl-D-aspartate) receptors of the nervous system, has an anti-inflammatory effect by reducing the concentration of IL-6 (interleukin 6) and tumor necrosis factor alpha. In adult patients, the need for morphine in the perioperative period is reduced when magnesium infusion is used. In current guidelines for treatment of acute pain in children, magnesium sulfate may be considered as a co-analgetic. However, the strength of such a recommendation is low due to the lack of reliable scientific research confirming the effectiveness of magnesium infusion in the pediatric population. The aim of this study is to evaluate the efficacy of intravenous magnesium sulfate infusion on the opioid consumption, the circulatory, metabolic and hormonal response to intubation and surgical trauma during anesthesia for laparoscopic appendectomy in children.

DETAILED DESCRIPTION:
Pain in the perioperative period is associated with surgical stimuli but also with laryngoscopy and intubation. According to the currently applicable ERAS (Enhanced Recovery After Surgery) doctrine, the recommended method of anesthesia is multimodal, low-opioid anesthesia. The essence of multimodal anesthesia is to combine different methods (e.g. general and regional anesthesia) and various anesthetic drugs in order to reduce the intraoperative use of opioids. The one of commonly used co-analgetic is magnesium. The use of magnesium infusion before induction of anesthesia may enhance the analgesic effect of the opioid administered before intubation. In current guidelines for the relief of acute pain in children, magnesium sulfate may be considered as a coanalgesic. It is based only on expert consensus opinion and/or data from small studies, retrospective studies, registries.

According to available data magnesium sulfate is superior to placebo in decreasing analgesic consumption and pain scores during the first 48 h after operation without any adverse effects in children with cerebral pals. In other groups of pediatric patients, the effectiveness of magnesium as a co-analgetic has not been proven. High quality randomized controlled trials are still missing.

The primary outcome of this study is to assess opioid consumption during the laparoscopic appendectomy. Number of patients requiring rescue dose of opioids will be measured.

The secondary aim is to examine total intraoperative fentanyl consumption, fluctuations of heart rate and blood pressure, metabolic, hormonal and inflammatory response (glucose, cortisol and IL-6 concentrations) and occurrence of side effects that may result from magnesium intake (decrease in blood pressure, bradycardia or allergic reaction).

In the pediatric population, the optimal perioperative magnesium dosage is 50 mg/kg as a bolus followed by an infusion of 15 mg/kg/hour until the end of the operation.

The general aim of the study is to evaluate the analgesic efficacy of intravenous magnesium sulfate as an adjunct to standard general anesthesia (involving intravenous induction and opioid with sevoflurane maintenance) for intubation and surgical trauma during anesthesia for laparoscopic appendectomy in children.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status class 1E, 2E, 3E (E - emergency)
* Patients undergoing laparoscopic appendectomy

Exclusion Criteria:

* Allergy to the magnesium sulfate or the excipient
* Hypermagnesemia
* Renal failure (GFR <30 ml/min)
* Myasthenia gravis
* Preoperative atrioventricular block
* Hypotension
* The use of digitalis glycosides
* The use of oral anticoagulants
* ASA physical status class 4E or higher
* Chronic treatment with analgesics
* Legal guardians or patient refusal

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients requiring rescue dose of opioids. | From tracheal intubation through to postanesthesia care unit admission (10 minutes after extubation).
  Patients who experience a 20% increase in BP (Blood Pressure) or HR (Heart Rate) from baseline during surgery and the early post-extubation period will receive a bolus of fentanyl (1 mcg/kg) as rescue analgesia. The number of these patients will be compared between the groups.
  Baseline parameters will be recorded after premedication with an IV bolus of 0.05 mg/kg midazolam, just before intubation.

SECONDARY OUTCOMES:
The requirement for opioids during anesthesia | From operating theatre admission through to postanesthesia care unit admission (10 minutes after extubation).
  Total amount of fentanyl in micrograms per kilogram of body weight used during anesthesia (dose for induction of anesthesia + doses added during surgery and in the early post-extubation period).
Hemodynamic reaction to tracheal intubation | Pre-intubation - immediately after intubation.
  A change in arterial blood pressure of more than 20% from baseline will be noted, and the fractions of these patients in each group will be compared. Baseline parameters will be recorded after premedication with an IV bolus of 0.05 mg/kg midazolam, just before intubation.
Metabolic response to laparoscopic procedure | From 5 minutes after tracheal intubation until the end of surgery, defined as the completion of dressing application.
  Glucose [mg/dl] levels will be measured and compared before and after laparoscopic procedure.
  The first blood sample will be taken 5 minutes after tracheal intubation, before the skin incision. The second blood sample will be taken immediately after the end of surgery, at the time of dressing application.
Hormonal response to laparoscopic procedure | From 5 minutes after tracheal intubation until the end of surgery, defined as the completion of dressing application.
  Cortisol levels [mcg/dl] will be measured and compared before and after laparoscopic procedure.
  The first blood sample will be taken 5 minutes after tracheal intubation, before the skin incision. The second blood sample will be taken immediately after the end of surgery, at the time of dressing application.
Inflammatory response to laparoscopic procedure | From 5 minutes after tracheal intubation until the end of surgery, defined as the completion of dressing application.
  IL-6 levels [pg/ml] will be measured and compared before and after laparoscopic procedure.
  The first blood sample will be taken 5 minutes after tracheal intubation, before the skin incision. The second blood sample will be taken immediately after the end of surgery, at the time of dressing application.
Magnesium blood level | From 5 minutes after tracheal intubation until the end of surgery, defined as the completion of dressing application.
  Magnesium level [mg/dl] will be measured after initial bolus and just before the end of its infusion.
  The first blood sample will be taken 5 minutes after tracheal intubation, before the skin incision. The second blood sample will be taken immediately after the end of surgery, at the time of dressing application. Magnesium infusion will be discontinued after the second blood sample is collected.
Side effects of magnesium sulfate | From the beginning of magnesium sulfate application until transfer to the postanesthesia care unit (10 minutes after extubation).
  Side effects of magnesium sulfate will be assessed by recording the rates of the following complications: hypotension & bradycardia (both defined as 2 SD (standard deviation) below the 50th percentile for age), allergic reaction. Need to discontinue the magnesium sulfate/placebo infusion due to side effects.
  Need to administer calcium gluconate.

OTHER OUTCOMES:
Length of stay in the hospital after completing anesthesia | From the time of extubation until the time of discharge from the hospital, through study completion, an average of 3 days.
  Length of stay in the hospital after completing anesthesia is defined as the time period from extubation (endotracheal tube removal) to discharge from the hospital. The mean length of hospital stay in the control and study groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Izabela Pągowska-Klimek, prof., Study Director — Medical University of Warsaw
Locations (1):
- Uniwersity Clinic Centre of Medical Uniwersity of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: The study protocol will be available to other researchers continuously after its publication.
  The Clinical Study Report will be published after the study completion.
Access Criteria: The datasets used and/or analysed during the study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Cettler M, Zielinska M, Rosada-Kurasinska J, Kubica-Cielinska A, Jarosz K, Bartkowska-Sniatkowska A. Guidelines for treatment of acute pain in children - the consensus statement of the Section of Paediatric Anaesthesiology and Intensive Therapy of the Polish Society of Anaesthesiology and Intensive Therapy. Anaesthesiol Intensive Ther. 2022;54(3):197-218. doi: 10.5114/ait.2022.118972. PMID 36189904
- [Background] Benzon HA, Shah RD, Hansen J, Hajduk J, Billings KR, De Oliveira GS Jr, Suresh S. The Effect of Systemic Magnesium on Postsurgical Pain in Children Undergoing Tonsillectomies: A Double-Blinded, Randomized, Placebo-Controlled Trial. Anesth Analg. 2015 Dec;121(6):1627-31. doi: 10.1213/ANE.0000000000001028. PMID 26501831
- [Background] O'Flaherty JE, Lin CX. Does ketamine or magnesium affect posttonsillectomy pain in children? Paediatr Anaesth. 2003 Jun;13(5):413-21. doi: 10.1046/j.1460-9592.2003.01049.x. PMID 12791115